CLINICAL TRIAL: NCT02983448
Title: Noninvasive Neuromodulation to Reserve Diastolic Dysfunction
Acronym: NERDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Stavros Stavrakis, Assistant Professor, University of Oklahoma
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-7147
Record Dates: First submitted 2016-11-30; First posted 2016-12-06 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure, Diastolic
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham stimulation first (Placebo Comparator): Sham stimulation delivered at the earlobe (devoid of vagal innervation) is given on first session.
  Transcutaneous vagus nerve stimulation delivered at the tragus (vagal innervation) is given on second session.
  Interventions: Device: transcutaneous vagus nerve stimulation
- Active stimulation first (Active Comparator): Transcutaneous vagus nerve stimulation delivered at the earlobe (vagal innervation) is given on first session.
  Sham stimulation delivered at the tragus (devoid of vagal innervation) is given on second session.
  Interventions: Device: transcutaneous vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation — All patients will receive both active and sham transcutaneous vagus nerve stimulation, with the order being randomized

SUMMARY:
This is a 2x2 cross over pilot study using low level transcutaneous vagus nerve stimulation (LLTS) to reverse diastolic dysfunction in patients with diastolic dysfunction. All patients will receive 2 separate, 1-hour sequences, at least 1 day apart, of active and sham LLTS, but the sequence will be randomized. Patients will be randomly assigned (1:1) to active/sham or sham/active LLTS. LLTS will be performed using a transcutaneous electrical nerve stimulation (TENS) device with electrodes attached to the tragus of the ear, which is innervated by auricular branch of the vagus nerve. Echocardiography will be performed after 30 minutes of LLTS or sham stimulation to assess diastolic function. Five-minute ECGs will be obtained for HRV analysis every 15 minutes of stimulation (total of 4 recordings).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients older than 18 year old
2. Evidence of diastolic dysfunction on echocardiogram within 24 months of study enrollment

Exclusion Criteria:

1. Left ventricular dysfunction (Left ventricular ejection fraction <40%)
2. Significant valvular disorder (i.e., prosthetic valve or hemodynamically relevant valvular diseases)
3. Recent (<6 months) stroke or myocardial infarction
4. Severe heart failure (NYHA class III or IV)
5. Recurrent vaso-vagal syncopal episodes
6. Unilateral or bilateral vagotomy
7. Pregnancy or breast feeding
8. Sick sinus syndrome (without a pacemaker), 2nd or 3rd degree AV block, bifascicular block or prolonged (PR>300ms) 1st degree AV block

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tran N, Asad Z, Elkholey K, Scherlag BJ, Po SS, Stavrakis S. Autonomic Neuromodulation Acutely Ameliorates Left Ventricular Strain in Humans. J Cardiovasc Transl Res. 2019 Jun;12(3):221-230. doi: 10.1007/s12265-018-9853-6. Epub 2018 Dec 17. PMID 30560316

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Stimulation First: Sham stimulation delivered at the earlobe (devoid of vagal innervation) is given on first session.
  Transcutaneous vagus nerve stimulation delivered at the tragus (vagal innervation) is given on second session.
  transcutaneous vagus nerve stimulation: All patients will receive both active and sham transcutaneous vagus nerve stimulation, with the order being randomized
- Active Stimulation First: Transcutaneous vagus nerve stimulation delivered at the earlobe (vagal innervation) is given on first session.
  Sham stimulation delivered at the tragus (devoid of vagal innervation) is given on second session.
  transcutaneous vagus nerve stimulation: All patients will receive both active and sham transcutaneous vagus nerve stimulation, with the order being randomized
Period: Overall Study
Arm/Group | Sham Stimulation First | Active Stimulation First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All patients will receive both active and sham transcutaneous vagus nerve stimulation, with the order being randomized
Arm/Group | All Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Echocardiographic Markers of Diastolic Dysfunction
Description: Global longitudinal strain
Time Frame: after 1 hour of stimulation
Population: All patients received both active and sham transcutaneous vagus nerve stimulation, with the order being randomized. The comparison is between active and sham stimulation.
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Sham Stimulation: Sham stimulation delivered at the earlobe (devoid of vagal innervation) is given on first session.
  Transcutaneous vagus nerve stimulation delivered at the tragus (vagal innervation) is given on second session.
  transcutaneous vagus nerve stimulation: All patients will receive both active and sham transcutaneous vagus nerve stimulation, with the order being randomized
- Active Stimulation: Transcutaneous vagus nerve stimulation delivered at the earlobe (vagal innervation) is given on first session.
  Sham stimulation delivered at the tragus (devoid of vagal innervation) is given on second session.
  transcutaneous vagus nerve stimulation: All patients will receive both active and sham transcutaneous vagus nerve stimulation, with the order being randomized
Arm/Group | Sham Stimulation | Active Stimulation
Number analyzed (Participants) | 24 | 24
percent | -21.2 (3) | -23.0 (2.8)

2. Secondary Outcome: Heart Rate Variability Measures
Description: low frequency to high frequency ratio. This is a measure of sympathovagal balance. A lower value reflects a more favorable balance between sympathetic and parasympathetic (vagal) tone.
Time Frame: after 1 hour of stimulation
Population: All patients will receive both active and sham transcutaneous vagus nerve stimulation, with the order being randomized. The comparison is between active and sham stimulation.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Sham Stimulation; Active Stimulation: All patients will receive both active and sham transcutaneous vagus nerve stimulation, with the order being randomized
Arm/Group | Sham Stimulation | Active Stimulation
Number analyzed (Participants) | 24 | 24
ratio | 3.1 (0.4) | 1.8 (0.4)

ADVERSE EVENTS:
Time Frame: through study completion (1 week)
Groups:
- Sham Intervention; Active Intervention: Transcutaneous vagus nerve stimulation delivered at the earlobe (vagal innervation) is given on first session.
  Sham stimulation delivered at the tragus (devoid of vagal innervation) is given on second session.
  transcutaneous vagus nerve stimulation: All patients will receive both active and sham transcutaneous vagus nerve stimulation, with the order being randomized
Arm/Group | Sham Intervention | Active Intervention
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT02983448/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT02983448/Prot_SAP_001.pdf